CLINICAL TRIAL: NCT05397418
Title: Effectiveness of a 12-week Low Impact Resistance Training Programme on Muscle Function, Body Composition, Quality of Life and Muscle Protein Synthesis in Women Aged 40-60 Years
Brief Title: Female Muscle Enhancement
Acronym: FemME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: P.volve LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2021-22-13; 309199 (Other: IRAS)
Record Dates: First submitted 2022-01-13; First posted 2022-05-31 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Muscle Function
Keywords: Muscle function; Females; Resistance exercise

STUDY DESIGN:
Intervention Model Description: Two-arm parallel unblinded randomised design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Supervised exercise program week 1-12, unsupervised exercise week 13-24.
  Interventions: Behavioral: Supervised resistance exercise program; Behavioral: Unsupervised resistance exercise program
- Control group (Sham Comparator): Maintain habitual activity week 1-12, unsupervised exercise week 13-24.
  Interventions: Behavioral: Unsupervised resistance exercise program

INTERVENTIONS:
Behavioral: Supervised resistance exercise program — 12 week supervised low impact resistance training program
  Arms: Intervention group
Behavioral: Unsupervised resistance exercise program — 12 week unsupervised low impact resistance training program

SUMMARY:
Participating in regular physical activity has been shown to reduce the risk of developing some diseases and disabilities that can occur with ageing. Muscles naturally decline with age, and in females this appears to occur more so around the time of menopause. Time, work, family commitments and the availability of facilities have all been identified as barriers to exercise in middle age.

Increasing activity levels in middle age appears to improve muscle function and bone health. However, there is a lack of evidence in how muscle function responds to low impact resistance exercise in middle aged females.

This study aims to assess the effectiveness and the mechanisms associated with building muscle as well as the effect on quality of life in middle aged (40-60 years) females using a low impact resistance training programme.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 40-60 years of age at time of screening.
* Body mass index <30kg/m2 and >18.5kg/m2
* Considered moderately active according to the 7 day International Physical Activity Questionnaire (IPAQ) (Craig et al., 2003)
* Self-reported as healthy (absence of injury or disease).
* Availability and willingness to attended 12 weeks of exercises classes 4-5 times per week at St Luke's Campus Exeter and participate in the study lasting a total of 26 weeks.

Exclusion Criteria:

* Pregnant, lactating or planning a pregnancy.
* Current diagnosis of a chronic disease such as diabetes, autoimmune disease, cardiovascular disease, kidney disease.
* Hysterectomy and/or ovariectomy.
* Currently prescribed hormone replacement therapy.
* Hypertension (BP ≥149/90 mm/Hg)
* Either current smoker, or history of smoking in the past 6 months.
* Currently taking supplements that have been shown to impact muscle function and muscle mass, such as creatine, in the last 6 months.
* Prescribed medications that have been shown to impact muscle function and muscle mass, such as steroids, in the last 6 months.
* History of epilepsy.
* Current or recent injury within the last 6 months that may affect their ability to carry out the resistance training program.
* Advised not to exercise by their General Practitioner or medical professional.
* Resistance training consistently for 3 or more times per week for the last 2 months

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2023-11-23 (Actual)

PRIMARY OUTCOMES:
Muscle function | 12 weeks
  Peak torque (Nm) of the shoulder and hip

SECONDARY OUTCOMES:
Body composition | 12 weeks
  Changes in fat mass and lean body mass
Bone mineral density | 12 weeks
  Changes in bone mineral density
Muscle thickness | 12 weeks
  Changes in muscle thickness
Muscle protein synthesis | 12 weeks
  Rate of muscle protein synthesis
Energy expenditure | 12 weeks
  Changes in energy expenditure rates
Sleep Quality | 12 weeks
  Changes in sleep quality using the Pittsburgh sleep quality index (PSQI) questionnaire
Self reported quality of life | 12 weeks
  Changes in self reported wellbeing measures using the Short Form Survey (SF-36)
Physical activity levels | 12 weeks
  Changes in physical activity energy expenditure as measured using an accelerometer
Exercise program acceptability | 12 weeks
  Changes in the rating of enjoyment of leisure time activity using the Groningen Enjoyment Questionnaire to rate enjoyment of exercise on a scale from strongly disagree to strongly agree
Changes in balance | 12 weeks
  Balance measured using the Y-balance test
Changes in flexibility | 12 weeks
  Flexibility measured using distance (cm) in zipper and sit and reach test
Changes in cardiovascular risk markers | 12 weeks
  Changes in biochemical lipid profile
Changes in diabetes risk markers | 12 weeks
  Changes in biochemical measures of HbA1c

OTHER OUTCOMES:
Sustainability of the exercise program through monitoring class attendance when unsupervised. | 12 weeks
  Suitability of the exercise program as a sustainable form of unsupervised online exercise as recorded in participant exercise diaries.

CONTACTS AND LOCATIONS:
Overall Officials: Francis Stephens, Principal Investigator — University of Exeter
Locations (1):
- University of Exeter, Exeter, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Svensen E, Koscien CP, Alamdari N, Wall BT, Stephens FB. A Novel Low-Impact Resistance Exercise Program Increases Strength and Balance in Females Irrespective of Menopause Status. Med Sci Sports Exerc. 2025 Mar 1;57(3):501-513. doi: 10.1249/MSS.0000000000003586. Epub 2024 Nov 6. PMID 39480197